CLINICAL TRIAL: NCT03386422
Title: "Pilot Study to Compare the Effectiveness of a Mindfulness Self-Compassion Intervention Versus a Cognitive-Behavioural Intervention to Improve Self-care and Quality of Life in a Chronic Pain Sample"
Brief Title: Mindfulness Self-Compassion Intervention Versus a Cognitive-Behavioral Intervention to Improve Self-care in Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Principal Investigator, Angela Palao, Psychiatry. PhD., Instituto de Investigación Hospital Universitario La Paz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1
Record Dates: First submitted 2017-12-08; First posted 2017-12-29 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Chronic Pain
Keywords: Mindfulness; Self-Compassion; Chronic Pain; Psychological Intervention; Cognitive-Behavioural therapy; acceptance; catastrophising; Self-Care; Quality of life
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Self-Compassion Intervention MSC (Experimental): Mindfulness Self-Compassion (MSC) is a standardized program to increase self-compassion. It has been developed by Neff and Germer. The structure of the program is similar to de Mindfulness-Based Stress Reduction program (MBSR), with duration of sessions between 2 and 2 hours and a half. The frequency of the sessions is one per week for 8 weeks, with practical and experiential exercices in sessions and between sessions.
  The MSC program focuses primary on helping patients to develop self-compassion, and it includes Mindfulness just as a secondary component.
  The MSC program will be conducted by a clinician trained in this specific program.
  Interventions: Behavioral: MSC
- Cognitive-Behavioural Intervention CBT (Active Comparator): It has been adapted a Cognitive-Behavioural Intervention for Chronic Pain by Moix and Kovacs. Our program will have 8 sessions, with duration of sessions between 2 and 2 hours and a half. The frequency of the sessions is one per week for 8 weeks, with homework between sessions.
  During these 8 sessions we will train the following techniques: psychoeducation about pain, relaxation training, cognitive restructuring training, solving problem training, psychoeducation about emotions, interpersonal skills and time organization.
  Interventions: Behavioral: CBT

INTERVENTIONS:
Behavioral: MSC — Mindfulness and Self-Compassion training
  Arms: Mindfulness Self-Compassion Intervention MSC
Behavioral: CBT — Cognitive-behavioural techniques training
  Arms: Cognitive-Behavioural Intervention CBT

SUMMARY:
Approximately 10-23% of people suffer from chronic pain in our country. Chronic pain is associated with emotional distress (anxiety and depression), physical and social impairment and reduction of quality of life in patients who suffer from this condition.

Self-Compassion is a useful attitude in order to regulate emotions, to be able to accept the experience that one is going through and to improve self-care in general population. Cognitive-behavioral programs (CBT) have already demonstrated that they are effective in order to reduce catastrophizing and passive coping with pain. However, effects of Mindful Self-Compassion interventions (based on mindfulness skills but not only) on chronic pain condition are still unknown.

The investigator's principal hypothesis is: MSC program will be, at least, as effective as CBT program in order to improve quality of life, self-compassion, self-care and acceptance capacity; and as effective as CBT to reduce catastrophizing, anxiety and depression in a chronic pain patients sample.

Moreover, investigators also hypothesize that MSC program will be, at least, as effective as CBT program in order to maintain the achieved benefits in a 6 months follow-up.

Investigators will conduct a Randomized Controlled Trial with two treatment arms in a chronic pain sample of patients of Hospital Universitario La Paz, Madrid.

After all recollection of data is done, investigators will conduct statistic analysis in order to accept or refuse our hypothesis.

DETAILED DESCRIPTION:
Approximately 10-23% of people suffer from chronic pain in our country. Chronic pain is associated with emotional distress (anxiety and depression), physical and social impairment and reduction of quality of life in patients who suffer from this condition.

Recent studies have elucidated that some conditions are clearly correlated with chronic pain, and could explain emotional distress and impairment in these patients. Such conditions are: attention bias to pain, cognitive inflexibility, fear avoidance, catastrophizing, passive coping with pain and no acceptance.

Recent meta-analysis suggest that Mindfulness-based interventions reduce anxiety and pain interference in daily life in patients with chronic pain. They do so through mechanisms that improve capacity of acceptance (whatever the experience is) and reduce catastrophizing. Self-Compassion is a useful attitude in order to regulate emotions, to be able to accept the experience that one is going through and to improve self-care in general population. Cognitive-behavioral programs (CBT) have already demonstrated that they are effective in order to reduce catastrophizing and passive coping with pain. However, effects of Mindful Self-Compassion interventions (based on mindfulness skills but not only) on chronic pain condition are still unknown.

Neff and Germer have developed a specific program to enhance self-compassion named Mindful Self-Compassion (MSC) that could be helpful to people with clinical problems. In spite of promising results of this interventions based on acceptation and self-compassion, its effectiveness on chronic pain conditions remains still unclear.

Investigator's principal hypothesis is: MSC program will be, at least, as effective as CBT program in order to improve quality of life, self-compassion, self-care and acceptance capacity; and as effective as CBT to reduce catastrophizing, anxiety and depression in a chronic pain patients sample.

Moreover, investigators also hypothesize that MSC program will be, at least, as effective as CBT program in order to maintain the achieved benefits in a 6 months follow-up.

Investigators will conduct a Randomized Controlled Trial with two treatment arms in a chronic pain sample of patients of Hospital Universitario La Paz, Madrid.

Both interventions will have 8 sessions, weekly frequency, duration of 2 hours and a half per session, and both programs will be conducted by clinical experts.

Investigators will asses levels of anxiety, depression, catastrophizing, pain interference, pain intensity, self-compassion and quality of life at the beginning of the intervention, at the end of the intervention, and a 6 months follow-up. Investigators also will administer a socio-demographic questionnaire at the beginning of the intervention to collect data about age, gender and pain characteristics.

After all recollection of data is done, investigators will conduct statistic analysis in order to accept or refuse their hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years old.
* Being in treatment in the Chronic Pain Unit at Hospital Universitario La Paz because of having a chronic pain of more than 3 months of duration, no matter the aetiology.
* Capable of understanding and giving his or her written informed consent.
* Significant levels of distress related to the pain at the beginning of treatment, assessed by clinical interview and HADS (HADS-A or HADS-D > or = 8).
* Patients that meet criteria for Mixed Adaptive Disorder, mild to moderate Depressive Disorder or Dysthymia, assessed by clinical interview conducted by a psychiatry of the Chronic Pain Unit or Mental Health Center.

Exclusion Criteria:

* Intelectual disability or cognitive impairment or dementia.
* Insufficient knowledge of the language to understand and participate on the intervention program.
* Serious mental illness in acute state at the moment of the beginning of the intervention.
* Substance abuse in the last 6 months.
* Autolytic ideas at the moment of the assessment.
* Previous training in mindfulness or CBT techniques.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2017-02-03 (Actual); Primary Completion 2018-12-07 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Self-Compassion | Up to 8 weeks
  Self-Compassion Scale (SCS, long version). Self-compassion and Self-care. Self-kindness, Common Humanity and Mindfulness. 26 items. Total score and 3 sub-scores from 1 to 5. Likert scale from 1 to 5.

SECONDARY OUTCOMES:
Acceptance | Up to 8 weeks
  Chronic Pain Acceptance Questionnaire (CPAQ). 2 factors: Activity engagement and Pain willingness.
Acceptance | In a 6 months follow-up
  Chronic Pain Acceptance Questionnaire (CPAQ). 2 factors: Activity engagement and Pain willingness.
Acceptance | Day 1 of the intervention
  Chronic Pain Acceptance Questionnaire (CPAQ). 2 factors: Activity engagement and Pain willingness.
Pain Interference | Up to 8 weeks
  Pain interference in daily life. Brief Pain Inventory (BPI): pain intensity and impact of pain in daily life. Investigators will use Impact in daily life sub-scale (7 items). Scores are from 0 to10.
Pain Interference | In a 6 months follow-up
  Pain interference in daily life. Brief Pain Inventory (BPI): pain intensity and impact of pain in daily life. Investigators will use Impact in daily life sub-scale (7 items). Scores are from 0 to10.
Pain Interference | Day 1 of the intervention
  Pain interference in daily life. Brief Pain Inventory (BPI): pain intensity and impact of pain in daily life. Investigators will use Impact in daily life sub-scale (7 items). Scores are from 0 to10.
Pain Intensity | Up to 8 weeks.
  Analogical Visual Scale. From 0 to 10 scores.
Pain Intensity | In a 6 months follow-up
  Analogical Visual Scale. From 0 to 10 scores.
Pain Intensity | Day 1 of the intervention
  Analogical Visual Scale. From 0 to 10 scores.
Catastrophising | Up to 8 weeks.
  Pain Catastrophising Scale (PCS). Rumination, magnification of consequences and hopelessness. 13 items, self-administered.
Catastrophising | In a 6 months follow-up
  Pain Catastrophising Scale (PCS). Rumination, magnification of consequences and hopelessness. 13 items, self-administered.
Catastrophising | Day 1 of the intervention
  Pain Catastrophising Scale (PCS). Rumination, magnification of consequences and hopelessness. 13 items, self-administered.
Quality of life | Up to 8 weeks.
  Health-Related Quality Of Life, Short Form (SF-36). 36 items. 8 sub-scores, no total score. Physical function, physical role, body pain, general state of health, vitality, social function, emotional role and mental health.
Quality of life | In a 6 months follow-up
  Health-Related Quality Of Life, Short Form (SF-36). 36 items. 8 sub-scores, no total score. Physical function, physical role, body pain, general state of health, vitality, social function, emotional role and mental health.
Quality of life | Day 1 of the intervention
  Health-Related Quality Of Life, Short Form (SF-36). 36 items. 8 sub-scores, no total score. Physical function, physical role, body pain, general state of health, vitality, social function, emotional role and mental health.
Anxiety and Depression | Up to 8 weeks.
  Levels of anxiety and depression. Symptomatology. Hospital Anxiety and Depression Scale (HADS). 14 items. 2 separated scores, 7 items each: anxiety and depression.
Anxiety and Depression | In a 6 months follow-up
  Levels of anxiety and depression. Symptomatology. Hospital Anxiety and Depression Scale (HADS). 14 items. 2 separated scores, 7 items each: anxiety and depression.
Anxiety and Depression | Day 1 of the intervention
  Levels of anxiety and depression. Symptomatology. Hospital Anxiety and Depression Scale (HADS). 14 items. 2 separated scores, 7 items each: anxiety and depression.
Satisfaction with the treatment | Up to 8 weeks.
  Satisfaction with the treatment (CRES-4). 4 questions. Scores from 0 to 300. The higher the punctuation, the higher satisfaction with treatment.
Adherence to the treatment | Up to 8 weeks.
  Adherence to the treatment (Number of sessions that one patient attends)
Self-Compassion | In a 6 months follow-up
  Self-Compassion Scale (SCS, long version). Self-compassion and Self-care. Self-kindness, Common Humanity and Mindfulness. 26 items. Total score and 3 sub-scores from 1 to 5. Likert scale from 1 to 5.
Self-Compassion | Day 1 of the intervention
  Self-Compassion Scale (SCS, long version). Self-compassion and Self-care. Self-kindness, Common Humanity and Mindfulness. 26 items. Total score and 3 sub-scores from 1 to 5. Likert scale from 1 to 5.

OTHER OUTCOMES:
Socio- demographic Data: Number of visited doctors. | Day 1 of the intervention
  Number of visited doctors in the last 3 months. Sociodemographic data Questionnaire.
Socio- demographic Data: Number of visits to emergency units. | Day 1 of the intervention
  Number of visits to emergency units in the last 3 months. Sociodemographic data Questionnaire.
Socio- demographic Data: course of pain expectation. | Day 1 of the intervention
  Course of pain that the patient expects (improvement, same condition, progressive worsening…) at the moment the intervention starts. Socio-demographic data Questionnaire.
Socio- demographic Data: psychiatric history. | Day 1 of the intervention
  Psychiatric history: whether the patient has or has not a history of mental health services visits for some kind of mental disorder. Socio-demographic data questionnaire.
Socio- demographic Data: type of pain. | Day 1 of the intervention
  Type of pain: area of pain in the body, diagnosis related to pain made for patient's doctor. Socio-demographic data Questionnaire.
Socio- demographic Data: time since pain started. | Day 1 of the intervention
  Time since the pain started: amount of time the patient has lived with pain. Socio-demographic data Questionnaire.
Socio- demographic Data: job status. | Day 1 of the intervention
  Job status: whether the patient is student, employed, unemployed, retired, or has a pension because of his/her disability. Socio-demographic data Questionnaire.
Socio- demographic Data: family life. | Day 1 of the intervention
  Family life: It is asked with whom the patient lives (couple, alone, kids, kids and couple…), if he/she has kids and if he/she lives with them. Socio-demographic data Questionnaire.
Socio- demographic Data: Marital Status | Day 1 of the intervention
  Marital Status: whether the patient is single, married or in a couple, divorced, or widower. Socio-demographic data Questionnaire.
Socio- demographic Data: Gender | Day 1 of the intervention
  Gender: Male or female. Socio-demographic data Questionnaire.
Socio- demographic Data: Age | Day 1 of the intervention
  Age of the patient. Socio-demographic data Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz Rodríguez Vega, Study Director — Hospital Universitario La Paz. Universidad Autónoma de Madrid.
Locations (1):
- Hospital Universitario La Paz., Madrid, Spain